CLINICAL TRIAL: NCT00648115
Title: Evaluating Vocational Materials for Incarcerated Veterans With Mental Illness
Brief Title: Evaluating Vocational Materials for Incarcerated Veterans With Mental Illness or Substance Abuse
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: D6192-R; 08-004 (Other: VANTHCS IRB)
Record Dates: First submitted 2008-03-27; First posted 2008-04-01 (Estimated); Results first posted 2015-10-30 (Estimated); Last update posted 2017-12-18 (Actual); Status verified 2017-11

CONDITIONS: Mental Illness
Keywords: Veterans; Substance-Related Disorders; Mental Health
MeSH Terms: conditions — Mental Disorders; Substance-Related Disorders; Psychological Well-Being

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Basic Vocational Services (Other): Veteran receives basic vocational services
  Interventions: Other: Basic Vocational Services
- Self-Study (Active Comparator): Veteran participates in self-study vocational program
  Interventions: Other: Self-Study
- Group program (Active Comparator): Group based vocational program
  Interventions: Other: Group Program

INTERVENTIONS:
Other: Basic Vocational Services — Vocational services
  Arms: Basic Vocational Services
Other: Self-Study — Veteran receives self-study resources
  Arms: Self-Study
Other: Group Program — Veteran participates in group vocational program
  Arms: Group program

SUMMARY:
The purpose of this research is to test the usefulness of a vocational rehabilitation program for veterans with a history of felonies who also have a mental illness or have substance dependency.

DETAILED DESCRIPTION:
The Department of Justice's Bureau of Justice Statistics (BOJS, 2000) reported in 2000 over 225,000 veterans were incarcerated in the nations' criminal facilities; 1 in 5 of these veterans saw combat during service. Approximately 78,000 veterans annually will be released from incarceration with 30% of those released from incarceration are re-arrested within 3 months, 44.1% re-arrested at one year, and 67.5% within 3 years. These numbers are higher with those with serious mental illnesses: 54.3% re-arrest rates at one year and 72% at 3 years.

The living status that many of these veterans with felonies return to is dire. In a survey of dually diagnosed and mentally ill offenders, 22% of mentally ill offenders and 43% of mentally ill offenders with substance addiction believed they would be homeless upon release. Ex-felons often return to more disadvantaged communities where employment is scarce (La Vigne, Mamalian, Travis, & Visher, 2003). Employers are reluctant to hire those with a history of incarceration due to biases against ex-offenders or due to legal liability (Connerley, Arvey, & Bernardy, 2001) or other biases (Holzer, 1996). Overall, employers have been shown to be less likely to hire ex-convicts than those with little work experience or those who are receiving welfare benefits (Holtzer, 1996).

The goal of this study is to identify successful vocational re-integration modalities for mental health and/or substance dependent veterans recently released from incarceration and those with felony histories. Specific Goals are 1) test time to employment between manual conditions; 2) test total time employed over the 12 months following training period; and 3) test economic impact between manual conditions The study will be a controlled 3 group randomized design. The independent variable will be the amount of vocational services received. Veterans will be randomly assigned to one of three conditions: 1) Basic vocational services but no manualized vocational program; 2) self-study of the manualized program; and 3) a full program consisting of the manualized program with vocational staff and peer vocational support specialists. All veterans enrolled in the study will have access to a Veteran's Employment Resource Center to provide infrastructure for job search.

Three primary dependent variables will be used. The first is the time till employment. The second is the total time employed during the 12 months following training. The third will be the economic impact of the training through differences in services required (e.g. emergency room visits, food stamps, cost of shelters, costs of rearrests) and income earned. Type of job skills, job history, and time incarcerated are some of the variables that potentially will be statistically controlled.

ELIGIBILITY:
Inclusion Criteria:

* underemployed or unemployed
* has a mental health or substance dependence diagnosis
* desires to enter the workforce through competitive employment.
* History of at least one felony conviction

Emphasis will be placed on returning OEF/OIF veterans, combat veterans, and women veterans. Veterans entering the study can be recruited regardless of living situation.

Exclusion Criteria:

* pursuing disability benefits due to unemployability
* diagnosis of dementia or evidence of severe cognitive impairment
* impaired reality testing due to psychosis
* actively suicidal or homicidal.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 111 (Actual)
Dates: Start 2009-06-01 (Actual); Primary Completion 2014-10-01 (Actual); Study Completion 2017-09-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: James P. LePage, PhD, Principal Investigator — VA North Texas Health Care System Dallas VA Medical Center, Dallas, TX
Locations (1):
- VA North Texas Health Care System Dallas VA Medical Center, Dallas, TX, Dallas, Texas, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Garcia-Rea E, LePage JP. Reliability and validity of World Health Organization Quality of Life-100 in homeless substance-dependent veteran population. J Rehabil Res Dev. 2008;45(4):619-25. doi: 10.1682/jrrd.2007.03.0048. PMID 18712647
- [Result] LePage JP, Washington EL, Lewis AA, Johnson KE, Garcia-Rea EA. Effects of structured vocational services on job-search success in ex-offender veterans with mental illness: 3-month follow-up. J Rehabil Res Dev. 2011;48(3):277-86. doi: 10.1682/jrrd.2010.03.0032. PMID 21480102
- [Result] LePage JP, Lewis AA, Washington EL, Davis B, Glasgow A. Effects of structured vocational services in ex-offender veterans with mental illness: 6-month follow-up. J Rehabil Res Dev. 2013;50(2):183-92. doi: 10.1682/jrrd.2011.09.0163. PMID 23760999

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Veterans recruited throughout medical center
Pre-assignment Details: Veterans must have completed a one week follow-up after enrollment to be randomized and included in the analyses.
Groups:
- Basic Vocational Services: Basic vocational services but no manualized vocational program
- Self-Study: Self-study of vocational materials
  comparison of vocational programs: Veterans will be randomly assigned to one of three conditions: 1) Basic vocational services but no manualized vocational program; 2) a self-study of the manualized program materials; and 3) a full program consisting of the manualized program with vocational staff and peer vocational support specialists. All veterans enrolled in the study will have access to a Veteran's Employment Resource Center to provide infrastructure for job search.
- Group Program: a full program consisting of the manualized program with vocational staff and peer vocational support specialists
  comparison of vocational programs: Veterans will be randomly assigned to one of three conditions: 1) Basic vocational services but no manualized vocational program; 2) a self-study of the manualized program materials; and 3) a full program consisting of the manualized program with vocational staff and peer vocational support specialists. All veterans enrolled in the study will have access to a Veteran's Employment Resource Center to provide infrastructure for job search.
Period: Overall Study
Arm/Group | Basic Vocational Services | Self-Study | Group Program
Started | 42 | 42 | 27
Completed | 42 | 42 | 27
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Basic Vocational Services | Self-Study | Group Program | Total
Number analyzed (Participants) | 42 | 42 | 27 | 111
Age, Continuous [Mean (Standard Deviation); unit: years] | 51.4 (4.7) | 50.4 (4.5) | 51.2 (5.3) | 51.0 (4.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 0 | 2 | 3
  Male | 41 | 42 | 25 | 108
Race/Ethnicity, Customized [Number; unit: participants]
  Racial/Ethnic Minority | 39 | 38 | 24 | 101
  White/Non-Minority | 3 | 4 | 3 | 10
Region of Enrollment [Number; unit: participants]
  United States | 42 | 42 | 27 | 111

OUTCOME MEASURES:

1. Primary Outcome: Time Till Employment in Days
Description: Number of days until first day of competitive employment
Time Frame: 12 months
Measure: Mean (95% Confidence Interval); unit: number of days to first employment
Arm/Group | Basic Vocational Services | Self-Study | Group Program
Number analyzed (Participants) | 42 | 42 | 27
number of days to first employment | 308 [277 to 341] | 301 [277 to 343] | 214 [153 to 275]
Statistical Analysis 1: Comparison: Basic Vocational Services vs Self-Study vs Group Program; Test type: Superiority or Other; p < 0.05, Chi-squared; Pearson chi square = 7.3

2. Secondary Outcome: Test Economic Impact Between Manual Conditions (e.g., Cost-benefit Ratio)
Description: overall economic impact, in dollars, will be evaluated by the following formula: income - healthcare cost - cost of incarceration
Time Frame: 12 months
Measure: Mean (Standard Deviation); unit: dollars
Arm/Group | Basic Vocational Services | Self-Study | Group Program
Number analyzed (Participants) | 42 | 42 | 27
dollars | 944 (3548) | 304 (1549) | 4698 (11620)

ADVERSE EVENTS:
Groups:
- Arm 1: Basic vocational services but no manualized vocational program
- Arm 2: Self-study of vocational materials
  comparison of vocational programs: Veterans will be randomly assigned to one of three conditions: 1) Basic vocational services but no manualized vocational program; 2) a self-study of the manualized program materials; and 3) a full program consisting of the manualized program with vocational staff and peer vocational support specialists. All veterans enrolled in the study will have access to a Veteran's Employment Resource Center to provide infrastructure for job search.
- Arm 3: a full program consisting of the manualized program with vocational staff and peer vocational support specialists
  comparison of vocational programs: Veterans will be randomly assigned to one of three conditions: 1) Basic vocational services but no manualized vocational program; 2) a self-study of the manualized program materials; and 3) a full program consisting of the manualized program with vocational staff and peer vocational support specialists. All veterans enrolled in the study will have access to a Veteran's Employment Resource Center to provide infrastructure for job search.
Arm/Group | Arm 1 | Arm 2 | Arm 3
Serious Adverse Events (participants affected / at risk) | 0/42 | 0/42 | 0/27
Other Adverse Events (participants affected / at risk) | 0/42 | 0/42 | 0/27

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes